CLINICAL TRIAL: NCT01109407
Title: Natural History Study of Monoclonal Gammopathy of Undetermined Significance (MGUS) and Smoldering Myeloma (SMM)
Status: Terminated | Type: Observational
Why Stopped: PI Left before primary outcome was established
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100096; 10-C-0096
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Smoldering Myeloma; Monoclonal Gammopathy of Undetermined Significance
Keywords: Plasma Cell Neoplasm; Natural History; Translational Studies; Gene Expression Profiling; Protein Markers; Smoldering Myeloma; SMM; Monoclonal Gammopathy of Undetermined Significance; MGUS
MeSH Terms: conditions — Smoldering Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patients with MGUS or SMM: patients with either Monoclonal gammopathy of undetermined significance (MGUS) or smoldering myeloma (SMM)

SUMMARY:
Background:

- Multiple myeloma is a type of cancer that affects white blood cells and has a poor long-term survival rate. Two other types of cancer, monoclonal gammopathy of undetermined significance (MGUS) and smoldering myeloma (SMM), may eventually progress and develop into multiple myeloma. Researchers are interested in collecting samples from individuals who have been diagnosed with MGUS and SMM to study possible risk factors for developing multiple myeloma.

Objectives:

- To study risk factors that may cause MGUS and SMM to progress to multiple myeloma.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with either MGUS or SMM but do not have multiple myeloma.

Design:

* Participants will be examined by study researchers at the initial visit, at 6 months following enrollment, and every 12 months for a maximum of 5 years.
* The following tests may be performed: (1) blood and urine tests, (2) bone marrow aspiration and biopsy, (3) imaging studies, and (4) a skeletal survey (a series of skeletal X-rays of the skull, spine, pelvis, ribs, shoulders, upper arm, and thigh bones).
* Treatment will not be provided as part of this protocol. - Participants will remain on the study for 5 years, or until their MGUS or SMM progresses to multiple myeloma requiring treatment.

DETAILED DESCRIPTION:
Background:

* Multiple Myeloma (MM) is an incurable plasma cell neoplasm with a median survival of 3-4 years.
* Monoclonal gammopathy of undetermined significance (MGUS) and smoldering myeloma (SMM) are premalignant plasma cell proliferative disorders characterized by elevated monoclonal protein and bone marrow plasma cells. MGUS affects 3.2% of Caucasians over the age of 50 and has a 1% annual risk of progression to MM. approximately 3000 cases of SMM are diagnosed annually with a 10% annual risk of progression to MM.
* Current risk stratification schemes rely on serum protein markers and phenotyping by flow cytometry. While they can differentiate high and low risk patients, they cannot predict outcome for individual patients, are not integrated with one another, and have limited direct correlation to biology.
* Paired samples linked to clinical information can advance research into improved risk stratification, the pathogenesis of MGUS, SMM, and MM, and the potential for an early treatment window for these incurable diseases.

Objectives:

* To characterize the natural history and prognosis of MGUS and SMM
* To integrate protein markers (including immunoglobulin free light-chains) and immunophenotyping by flow cytometry with molecular profiles (including gene expression profiles) and clinical outcomes
* To apply expertise and diagnostic technology to provide improved evaluation, monitoring, and risk-stratification for patients on this protocol
* To provide paired samples of blood and tissue linked to clinical and molecular information for pilot translational studies

Eligibility:

* A confirmed diagnosis of MGUS or SMM (based on IMWG diagnostic criteria)
* Age greater than or equal to 18 years
* ECOG performance status in the range of 0-2
* Patients who have a diagnosis of MM are not eligible for this study.

Design:

* This is a prospective cohort study of patients with either MGUS or SMM.
* Following initial evaluation and confirmation of diagnosis, patients will be followed as clinically indicated, usually at 12 month intervals.
* The primary endpoint is progression to MM requiring treatment.
* Patients may donate cellular products or tissues as appropriate for research purposes.

  154 patients with MGUS and 154 patients with SMM will be enrolled on this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of MGUS and SMM will be made in accordance with the clinical diagnostic criteria set forth by the International Myeloma Working Group (Table 1).
* The diagnoses will be confirmed by either serum/urine protein electrophoresis, immunofixation and light-chain assays; or immunohistochemistry analyses of the bone marrow biopsy, or a combination of these tests.
* Age greater than or equal to 18 years.
* ECOG performance status of 0-2.
* The patient must be competent to sign an informed consent form.

EXCLUSION CRITERIA:

- A diagnosis of MM as defined as any patient with detectable M-protein in blood and/or urine, monoclonal plasma cells in the bone marrow, and evidence of end-organ damage (based on the International Myeloma Working Group s diagnostic CRAB criteria:

hypercalcemia [serum calcium at least 1 mg/dL above the upper limit of normal], renal failure [creatinine greater than 1.95 mg/dL), anemia (hemoglobin less than 10 g/dL], or bone lesions [lytic lesions or osteoporosis with compression fractures]).

- Patients who have received previous therapy for MM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MGUS or SMM will enroll on the study for the purpose of expert monitoring of their disease (MGUS or SMM), improved risk-stratification, and for the purpose of donating tissue and cellular products for research.@@@
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2010-04-22 (Actual); Primary Completion 2014-05-16 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Characterize the natural history and prognosis of MGUS and SMM | 6 months
  determination of subtypes of MM based on GEP, and determination of prognostic indicators
Integrate protein markers with molecular profiles and clinical outcomes. | 6 months
  comparison of molecular profiles and rate of disease progression per MM subtype

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Roschewski, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kristinsson SY, Landgren O, Dickman PW, Derolf AR, Bjorkholm M. Patterns of survival in multiple myeloma: a population-based study of patients diagnosed in Sweden from 1973 to 2003. J Clin Oncol. 2007 May 20;25(15):1993-9. doi: 10.1200/JCO.2006.09.0100. Epub 2007 Apr 9. PMID 17420512
- [Background] Kumar SK, Rajkumar SV, Dispenzieri A, Lacy MQ, Hayman SR, Buadi FK, Zeldenrust SR, Dingli D, Russell SJ, Lust JA, Greipp PR, Kyle RA, Gertz MA. Improved survival in multiple myeloma and the impact of novel therapies. Blood. 2008 Mar 1;111(5):2516-20. doi: 10.1182/blood-2007-10-116129. Epub 2007 Nov 1. PMID 17975015
- [Background] Landgren O, Kyle RA, Pfeiffer RM, Katzmann JA, Caporaso NE, Hayes RB, Dispenzieri A, Kumar S, Clark RJ, Baris D, Hoover R, Rajkumar SV. Monoclonal gammopathy of undetermined significance (MGUS) consistently precedes multiple myeloma: a prospective study. Blood. 2009 May 28;113(22):5412-7. doi: 10.1182/blood-2008-12-194241. Epub 2009 Jan 29. PMID 19179464
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0096.html